CLINICAL TRIAL: NCT01868165
Title: Assessing the Impact of Calcium Channel Blockers on COGnitive Function in the Very Elderly (AI-COG)
Status: Completed | Type: Observational
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Other Study IDs: P40221
Record Dates: First submitted 2013-05-29; First posted 2013-06-04 (Estimated); Results first posted 2019-09-23 (Actual); Last update posted 2019-09-23 (Actual); Status verified 2019-08

CONDITIONS: Cognitive Ability, General; High Blood Pressure
Keywords: Cognitive decline; High blood pressure; Hypertension; Ageing; Dementia; Antihypertensives
MeSH Terms: conditions — Hypertension; Cognitive Dysfunction; Dementia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Cohort of older adults taking antihypertensives: Adults aged 80 and over treated with antihypertensive drugs

SUMMARY:
Older adults are at increased risk of high blood pressure and cognitive decline. High blood pressure itself also increases risk of cognitive decline. A particular type of blood pressure lowering drug (a calcium channel blocker(CCB)) may lower risk of dementia in younger adults but there is no clear evidence of it's impact in those >=80. It is important that we know whether CCB use impacts on cognitive function in this age group. This study will examine the impact of antihypertensives on change in cognitive function with a particular focus on CCBs.

DETAILED DESCRIPTION:
This study is an observational cohort study examining cognitive change in those participants taking antihypertensives and aged 80 and over and examining cognitive change in participants taking different types of antihypertensive medication.

ELIGIBILITY:
Inclusion Criteria:

Aged 80 and over Receiving pharmacological treatment for hypertension Mini Mental State Exam score >24 No other condition likely to limit life to less than one year or to prevent the taking of informed consent.

Exclusion Criteria:

Aged under 80 years Not receiving pharmacological treatment for hypertension Mini Mental State Exam score <25 Diagnosed with a condition likely to limit life to less than one year or to prevent the taking of informed consent.

Presence of a sensory impairment or an existing neuropsychological deficit of sufficient severity to prevent cognitive testing.

Presence of a condition that will prevent cognitive testing, registered blind, profoundly deaf, suffering from an aphasia.

Min Age: 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: UK Primary care
Sampling Method: Non-Probability Sample
Enrollment: 337 (Actual)
Dates: Start 2013-06; Primary Completion 2015-02 (Actual); Study Completion 2016-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ruth Peters, PhD, Principal Investigator — Imperial College London, UK
Locations (7):
- United Kingdom (7):
  - The Kiltearn Medical Centre, Nantwich, Cheshire
  - Ashfields Primary Care Centre, Sandbach, Cheshire
  - Whitby Group Practice, Whitby, North Yorkshire
  - South Axholme Practice, Epworth, Yorkshire
  - Dr Moss and Partners, Harrogate
  - Gale Farm Surgery, York
  - Haxby Group Practice, York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Peters R. No clear relationship between antihypertensive class and cognitive function over 12 months in a cohort study of community-dwelling adults aged 80 and over. Ther Adv Chronic Dis. 2019 Jan 31;10:2040622318820849. doi: 10.1177/2040622318820849. eCollection 2019. PMID 30728929

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants had hypertension and treatment with antihypertensives.The study examined the cognitive change in older adults taking antihypertensives with a particular focus on Calcium Channel Blockers (CCB). Cognitive function was tested at 0 & 12 months. Participation in the study had no impact on treatment.
Groups:
- Older Adult Cohort: Older adults receiving treatment with antihypertensive medication
Period: Overall Study
Arm/Group | Older Adult Cohort
Started | 337
Completed | 292
Not Completed | 45
Not completed — Withdrawal by Subject | 36
Not completed — Physician Decision | 2
Not completed — Lost to Follow-up | 3
Not completed — Death | 4

BASELINE CHARACTERISTICS:
Arm/Group | Older Adult Cohort
Number analyzed (Participants) | 292
Age, Continuous [Mean (Standard Deviation); unit: years] | 83.5 (2.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 161
  Male | 131
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 288
  Asian | 1
  Black | 1
  Unspecified | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United Kingdom | 292
Extended Mini-Mental State Exam [Median (Inter-Quartile Range); unit: units on a scale] — The extended mini mental state exam is a widely used and validated cognitive screening tool. It is scored from 0-100 Higher values are better. A population without cognitive impairment would be expected to score near the maximum value.
  units on a scale | 95 [91 to 98]
Systolic blood pressure [Mean (Standard Deviation); unit: mmHg] | 137.1 (14.4)
Diastolic blood pressure [Mean (Standard Deviation); unit: mmHg] | 74.8 (9.7)
Prescribed calcium channel blockers [Count of Participants; unit: Participants] | 135
Cardiovascular disease [Count of Participants; unit: Participants] | 81
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 27.5 (4.5)

OUTCOME MEASURES:

1. Primary Outcome: Change in Cognitive Function as Measured Using the Extended Mini Mental State Exam
Description: The change in cognitive function measured using the extended mini-mental state exam (this is an extended screening test which assesses several areas of cognitive function, the scale is from 0-100, higher scores are better, those without cognitive impairment would be expected to score close to maximum)
Time Frame: 12 months
Population: Regression analysis examining change in cognitive function in older adults taking antihypertensives, results are reported for those taking calcium channel blocker antihypertensives over one year of follow up.
Measure: Mean (95% Confidence Interval); unit: Change on a scale
Groups:
- Older Adult Cohort: Older adult cohort receiving antihypertensive medication
Arm/Group | Older Adult Cohort
Number analyzed (Participants) | 292
Change on a scale | 0.58 [-0.60 to 1.77]
Statistical Analysis 1: Comparison: Older Adult Cohort; Test type: Other; Slope = 0.58, 95% CI 2-sided [-0.60 to 1.77] — Linear regression slope and 95% confidence intervals for the association between calcium channel blocker use and cognitive change was 0.58 (-0.60:1.77). Multiple adjustments including; age, sex, education

ADVERSE EVENTS:
Time Frame: 12 month
Groups:
- Older Adult Cohort: Older adults receiving antihypertensive medication
Arm/Group | Older Adult Cohort
All-Cause Mortality (participants affected / at risk) | 0/292
Serious Adverse Events (participants affected / at risk) | 0/292
Other Adverse Events (participants affected / at risk) | 0/292

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes